CLINICAL TRIAL: NCT03755895
Title: Randomized Trial Comparing the Hypnosis Versus Standard Care of Anxiety and Pain in Patients With Brachytherapy
Brief Title: Contribution of Hypnosis to Anxiety and Pain in Brachytherapy Patients
Acronym: HYCUDES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-004527-37
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Brachytherapy
Keywords: Cancer; hypnosis; care management
MeSH Terms: conditions — Neoplasms | interventions — kalinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental (Experimental): patients to benefit from brachytherapy detachment under KALINOX and formal hypnosis
  Interventions: Other: formal hypnosis; Drug: Kalinox
- active comparator (Active Comparator): patients to benefit from brachytherapy detachment under KALINOX
  Interventions: Drug: Kalinox

INTERVENTIONS:
Other: formal hypnosis — patients will have brachytherapy detachment under Kalinox and formal hypnosis
  Arms: experimental
Drug: Kalinox — patients will have brachytherapy detachment under Kalinox

SUMMARY:
Formal hypnosis is a non-drug technique known to decrease anxiety and pain during the preoperative procedure.

In brachytherapy, the practice of hypnosis has been shown to be feasible and beneficial for patients treated for prostate cancer The goal of the study is to demonstrate the added value of hypnosis during a brachytherapy detachment by improving the comfort of the patient.

The investigators want to evaluate the contribution of hypnosis during brachytherapy detachment by quantifying the anxiety and pain felt by the patient during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 and ≤ 80 years
* Patients expected to benefit a brachytherapy detachment Under KALINOX® for one of the types of applications described below:

  * Deep interstitial application: anal canal, vagina, vulva
  * Gynecological application: mold, Utrecht® system or Venezia® system
* Ability to provide written informed consent
* Patients affiliated to the social security system

Exclusion Criteria:

* Minor and patients over 80 years old
* Patients with major hearing loss
* Patients who had recent ocular surgery with oculiare gas injection.
* Patients suffering from psychotic disorders, and dementias.
* Patients who do not understand the French language
* Patients under guardianship or deprived of liberty
* Patients with a contraindication to the administration of KALINOX®

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluation | 1day
  The patient's anxiety will be assessed using the State-Trait Anxiety Inventory scale ("state of anxiety") before premedication (in the bedroom) and immediately after the brachytherapy detachment (in the examination room) during brachytherapy detachment using two care management: standard care versus standard care with formal hypnosis. The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety (Spielberger et al, 1983). The scale include 20 items. Higher scores indicate greater anxiety

SECONDARY OUTCOMES:
Pain evaluation: numeric scale | 1 day
  Pain will be evaluated by a numeric scale before premedication (in the room), just before and just after the brachytherapy detachment (in the examination room). Patient inform their level of pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain
Anxiety evaluation | 1 day
  Anxiety will be evaluated by a numeric scale just before and just after the brachytherapy detachment. Patient inform their level of anxiety from 0 to 10 (11 point scale) with the understanding that 0 is equal to no anxiety and 10 is equal to worst possible anxiety
Patient's perception of the care | 1day
  The patient's perception of the care will be evaluated by a semi-directive phone interview conducted by the medical staff between day 3 and day 5 after the brachytherapy detachment
Time of brachytherapy detachment | 1day
  The time of brachytherapy detachment will be noted from the entrance to the patient's examination room until the end of the brachytherapy detachment
Realization of the brachytherapy detachment | 1day
  The ease of realization of the brachytherapy detachment and the comfort of the medical staff will be evaluated by an numeric scale at the end of the care and by a self-survey

CONTACTS AND LOCATIONS:
Overall Officials: Sophie RENARD, Md, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemoine L, Adam V, Salleron J, Cuisinier C, Perrin J, Brunaud CC, Jean-Francois P, Bruand M, Peiffert D, Etienne R, Schohn CH, Renard S. Randomized trial comparing hypnosis versus standard management on patient anxiety and pain during pelvic brachytherapy applicator removal. Brachytherapy. 2025 Nov-Dec;24(6):854-862. doi: 10.1016/j.brachy.2025.07.010. Epub 2025 Aug 28. PMID 40883194